CLINICAL TRIAL: NCT05934396
Title: Practice Experiences for School Reintegration: An Immersive Virtual Reality Program to Enhance Skill Development of Hospitalized Adolescents
Brief Title: Practice Experiences for School Reintegration
Acronym: PrESR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20-3464; 5K23MH122775 (NIH)
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-01

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Enhanced Control (Active Comparator): Cognitive Behavioral Therapy (CBT) Worksheets
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets
- Affect Regulation (Active Comparator): Cognitive Behavioral Therapy (CBT) Worksheets; Safety Planning; Virtual Reality (VR) Enhanced Affect Regulation
  Interventions: Behavioral: Safety Planning; Behavioral: VR Enhanced Affect Regulation; Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets
- Problem Solving (Active Comparator): Cognitive Behavioral Therapy (CBT) Worksheets; Safety Planning; Virtual Reality (VR) Enhanced Problem Solving
  Interventions: Behavioral: Safety Planning; Behavioral: VR Enhanced Problem Solving; Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets
- Affect Regulation + Problem Solving (Active Comparator): Cognitive Behavioral Therapy (CBT) Worksheets; Safety Planning; Virtual Reality (VR) Enhanced Affect Regulation; VR Enhanced Problem Solving
  Interventions: Behavioral: Safety Planning; Behavioral: VR Enhanced Affect Regulation; Behavioral: VR Enhanced Problem Solving; Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets
- Cognitive Restructuring (Active Comparator): Cognitive Behavioral Therapy (CBT) Worksheets; Safety Planning; Virtual Reality (VR) Enhanced Cognitive Restructuring
  Interventions: Behavioral: Safety Planning; Behavioral: VR Enhanced Cognitive Restructuring; Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets
- Affect Regulation + Cognitive Restructuring (Active Comparator): Cognitive Behavioral Therapy (CBT) Worksheets; Safety Planning; Virtual Reality (VR) Enhanced Affect Regulation; VR Enhanced Cognitive Restructuring
  Interventions: Behavioral: Safety Planning; Behavioral: VR Enhanced Affect Regulation; Behavioral: VR Enhanced Cognitive Restructuring; Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets
- Cognitive Restructuring + Problem Solving (Active Comparator): Cognitive Behavioral Therapy (CBT) Worksheets; Safety Planning; Virtual Reality (VR) Enhanced Cognitive Restructuring; VR Enhanced Problem Solving
  Interventions: Behavioral: Safety Planning; Behavioral: VR Enhanced Cognitive Restructuring; Behavioral: VR Enhanced Problem Solving; Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets
- Affect Regulation + Cognitive Restructuring + Problem Solving (Active Comparator): Cognitive Behavioral Therapy (CBT) Worksheets; Safety Planning; Virtual Reality (VR) Enhanced Affect Regulation; VR Enhanced Cognitive Restructuring; VR Enhanced Problem Solving
  Interventions: Behavioral: Safety Planning; Behavioral: VR Enhanced Affect Regulation; Behavioral: VR Enhanced Cognitive Restructuring; Behavioral: VR Enhanced Problem Solving; Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets

INTERVENTIONS:
Behavioral: Safety Planning — Prior to discharge and following the conclusion of all Virtual Reality (VR) sessions, the participant will develop a safety planning intervention for school settings in collaboration with relevant individuals (e.g., the researcher, a school professional).
  Arms: Affect Regulation; Affect Regulation + Cognitive Restructuring; Affect Regulation + Cognitive Restructuring + Problem Solving; Affect Regulation + Problem Solving; Cognitive Restructuring; Cognitive Restructuring + Problem Solving; Problem Solving
Behavioral: VR Enhanced Affect Regulation — Participants will receive an overview of affect regulation in VR and then have the opportunity to practice using affect regulation in a brief immersive experience designed to mimic difficult school experiences. Each session begins with goal setting prior to the VR experience and concludes with a debrief summary following the VR experience.
  Arms: Affect Regulation; Affect Regulation + Cognitive Restructuring; Affect Regulation + Cognitive Restructuring + Problem Solving; Affect Regulation + Problem Solving
Behavioral: VR Enhanced Cognitive Restructuring — Participants will receive an overview of cognitive restructuring in VR and then have the opportunity to practice using cognitive restructuring in a brief immersive experience designed to mimic difficult school experiences. Each session begins with goal setting prior to the VR experience and concludes with a debrief summary following the VR experience.
  Arms: Affect Regulation + Cognitive Restructuring; Affect Regulation + Cognitive Restructuring + Problem Solving; Cognitive Restructuring; Cognitive Restructuring + Problem Solving
Behavioral: VR Enhanced Problem Solving — Participants will receive an overview of problem solving in VR and then have the opportunity to practice using problem solving in a brief immersive experience designed to mimic difficult school experiences. Each session begins with goal setting prior to the VR experience and concludes with a debrief summary following the VR experience.
  Arms: Affect Regulation + Cognitive Restructuring + Problem Solving; Affect Regulation + Problem Solving; Cognitive Restructuring + Problem Solving; Problem Solving
Behavioral: Cognitive Behavioral Therapy (CBT) Worksheets — The researchers will provide instructions for participants to complete a packet of worksheets teaching introduction to cognitive behavioral therapy (CBT), affect regulation, cognitive restructuring, and problem solving.

SUMMARY:
This study is developing and refining a novel Virtual Reality (VR) supplement for inpatient treatment: the Practice Experiences for School Reintegration (PrESR) program. The PrESR will provide immersive school experiences for inpatient adolescents (with suicidal-related admissions) to practice skills in real-world settings with the guidance of a trained clinician within the confines of a hospital. This pilot study follows a Multiphase Optimization Strategy (MOST) to conduct a pilot optimization trial of the PrESR to inform the feasibility of training clinicians, the ability to recruit adolescent inpatient participants, and management of experimental conditions. This study is not powered to test hypotheses; however, in addition to assessing feasibility and acceptability, this pilot trial will assess candidate intermediary and outcome measures.

DETAILED DESCRIPTION:
This study follows a multiphased optimization (MOST) research design; this clinical trial is considered to be a pilot optimization component of the MOST framework. For the present study, a prospective sample of adolescents hospitalized for suicidal thoughts and behaviors will be randomly selected into one of 8 experimental conditions (N=5-6 per group). Although the intervention for the pilot optimization trial will be implemented by a member of research staff, this study will also aim to recruit 2-5 clinicians to deliver the full intervention to a separate sample of adolescent patients to inform acceptability and feasibility of the intervention within their clinical workflow.

ELIGIBILITY:
Inclusion Criteria:

Adolescent Participants:

* current hospitalization for suicidal thoughts and behaviors
* ages 13-18
* expected return to school following discharge
* ability to speak, read, and understand English sufficiently to complete study procedures,
* consent of a parent/legal guardian (in English or Spanish; for minor participants)
* adolescent assent or consent (in English)
* clinician approval.

Hospital professionals:

* Works as a clinician at the hospital site who delivers treatment including CBT to hospitalized adolescents,
* Hospital professional consent (in English)
* consent of patient's parent/legal guardian (in English or Spanish; for minor participants)
* adolescent patient assent or consent (in English).

Exclusion Criteria:

Adolescent Participants

* evidence of active psychosis,
* evidence of intellectual disability
* Risk for Cyber-sickness (greater than or equal to 50th percentile as measured on the Motion Sickness Susceptibility Questionnaire)

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Marraccini, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Adolescent Psychiatry Inpatient Unit, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 125 parents/guardians were called based on chart review and 94 were successfully contacted; out of those, 54 provided permission for their adolescent to participate. Of 54 adolescents contacted, 48 provided assent, of whom 1 was screened out due to risk for cybersickness. Of the remaining 47 adolescents, 5 were in the open trial and 42 were in the optimization trial. 7 hospital professionals consented to participate in the open trial, of whom 4 delivered the intervention to at least one patient.
Groups:
- Affect Regulation + Cognitive Restructuring + Problem Solving: Cognitive Behavioral Therapy (CBT) Worksheets; Safety Planning; Virtual Reality (VR) Enhanced Affect Regulation; VR Enhanced Cognitive Restructuring; VR Enhanced Problem Solving
  Safety Planning: Prior to discharge and after Virtual Reality (VR) sessions, the participant develops a safety plan for schools.
  VR Enhanced Affect Regulation: Participants receive an overview of affect regulation in VR and then can practice using affect regulation in a brief immersive experience designed to mimic difficult school experiences. Each session begins with goal setting prior to the VR experience and concludes with a debrief summary.
  VR Enhanced Cognitive Restructuring: Participants receive an overview of cognitive restructuring in VR and then can practice using cognitive restructuring in a brief immersive experience designed to mimic difficult school experiences. Each session begins with goal setting prior to the VR experience and concludes with a debrief summary.
  VR Enhanced Problem Solving: Participants receive an overview of problem solving in VR and then can practice using problem solving in a brief immersive experience designed to mimic difficult school experiences. Each session begins with goal setting prior to the VR experience and concludes with a debrief summary.
  CBT Worksheets: The researchers will provide instructions for participants to complete a packet of worksheets teaching introduction to CBT, affect regulation, cognitive restructuring, and problem solving.
- Hospital Professionals: Clinicians who delivered the intervention to inform acceptability and feasibility of the intervention within their clinical workflow.
- Adolescent Patients Selected by Hospital Professionals: Adolescent patients receiving the intervention delivered by hospital professional participants
Period: Optimization Trial
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Started | 6 | 5 | 6 | 5 | 5 | 5 | 5 | 5 | 0 | 0
Completed Baseline | 6 | 5 | 6 | 4 | 5 | 5 | 4 | 5 | 0 | 0
Completed 2-Week Journal | 0 | 4 | 1 | 1 | 3 | 0 | 2 | 2 | 0 | 0
Completed 2-Week Return to School Follow-Up | 2 | 5 | 4 | 3 | 2 | 2 | 2 | 3 | 0 | 0
Completed 3-Month Return to School Follow-Up | 1 | 5 | 3 | 1 | 3 | 2 | 2 | 1 | 0 | 0
Completed | 0 | 4 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0
Not Completed | 6 | 1 | 5 | 5 | 3 | 5 | 3 | 4 | 0 | 0
Period: Open Trial Period
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Data pertaining to Adolescent Patients Selected by Hospital Professionals are only analyzed for the outcomes related to overall patient recruitment and screening: "Proportion of Patients in the Target Population Who Agree to Participate [Time Frame: Baseline]" and "Proportion of Patients in the Target Population Excluded Due to Motion Sickness Screening [Time Frame: Baseline]".
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals | Total
Number analyzed (Participants) | 6 | 5 | 6 | 5 | 5 | 5 | 5 | 5 | 7 | 5 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 6 | 5 | 5 | 5 | 5 | 5 | 0 | 5 | 47
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 7
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — For adolescents, sex/gender is categorized by sex (male, female, intersex) / gender (man/boy, woman/girl, in some other way, "I do not know what this question is asking", "I do not know if I am transgender"). For hospital professionals, sex/gender is categorized by sex (male, female) / gender (female, male, transgender, or "I do not identify as female, male, or transgender"). Unknown refers to missing data or not reported data.
  Participants
    Female/Girl/Woman | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 2 | 6 | 3 | 29
    Male/Boy/Man | 3 | 2 | 2 | 0 | 2 | 3 | 3 | 1 | 0 | 2 | 18
    Female/Identifies in Some Other Way | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
    Female/Boy/Man | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
    Unknown | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Female/Transgender | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 2 | 1 | 3 | 1 | 2 | 0 | 2 | 14
  Not Hispanic or Latino | 6 | 5 | 3 | 1 | 4 | 2 | 4 | 3 | 7 | 3 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 2 | 0 | 0 | 2 | 4 | 1 | 1 | 15
  White | 2 | 3 | 2 | 1 | 2 | 4 | 0 | 0 | 6 | 4 | 24
  More than one race | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 8
  Unknown or Not Reported | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 6 | 5 | 5 | 5 | 5 | 5 | 7 | 5 | 54

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in the Target Population Who Agree to Participate
Description: Recruitment rate was determined based on the proportion of adolescents providing assent and parents or legal guardians providing permission relative to the number of parents or legal guardians approached.
Time Frame: Baseline
Population: Analysis population includes adolescents hospitalized for suicide-related crises, identified through electronic health records and deemed appropriate for the intervention by clinicians, including those considered for the Optimization Trial and the Open Trial.
Measure: Number; unit: proportion of potential participants
Groups:
- All Potential Adolescent Participants Who Were Approached: Adolescents hospitalized for suicide-related crises, identified through electronic health records and deemed appropriate for the intervention by clinicians.
Arm/Group | All Potential Adolescent Participants Who Were Approached
Number analyzed (Participants) | 125
proportion of potential participants | 0.384

2. Primary Outcome: Proportion of Patients in the Target Population Excluded Due to Motion Sickness Screening
Description: Rate of recruitment related to motion sickness was determined based on the proportion of assented adolescents whose scores were >/= than 50th percentile on motion sickness questionnaire relative to the number of assented adolescents.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Groups:
- All Assented Adolescent Participants: Adolescents hospitalized for suicide-related crises who provided assent to participate in the study.
Arm/Group | All Assented Adolescent Participants
Number analyzed (Participants) | 48
proportion of participants | 0.021

3. Primary Outcome: Proportion of Participants Who Complete All Study Procedures
Description: Proportion of participants who complete all study procedures was determined based on the proportion of adolescents completing study procedures at Baseline, 2-week follow-up, 3-month follow-up, and journals over the two weeks of their return to school relative to the total number of adolescents participating in that condition.
Time Frame: up to 3-months following school re-entry
Population: This outcome applies to participants in the Optimization Trial only. Data were not collected for Hospital Professionals or Adolescent Patients Selected by Hospital Professionals for the Open Trial Period.
Measure: Number; unit: proportion of participants
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Number analyzed (Participants) | 6 | 5 | 6 | 5 | 5 | 5 | 5 | 5 | 0 | 0
proportion of participants | 0 | 0.800 | 0.167 | 0 | 0.400 | 0 | 0.400 | 0.200 |  |

4. Primary Outcome: Average Number of Hours to Complete Assessments at Each Time Point
Description: Time to complete assessments, assessments are expected to last less than 4 hours. Note that the number of participants to start a Period is not equal to the number who completed previous Period for "Affect Regulation + Problem Solving" and "Cognitive Restructuring + Problem Solving" because 1 participant in each condition was withdrawn or withdrew.
Time Frame: up to 3-months following school re-entry
Population: This outcome applies to participants in the Optimization Trial only. Data were not collected for Hospital Professionals or Adolescent Patients Selected by Hospital Professionals for the Open Trial Period. Numbers of Participants Analyzed per Row differs from the Overall Numbers of Participants due to number of individuals completing meetings across timepoints (i.e., not all participants completed every meeting).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Number analyzed (Participants) | 5 | 5 | 6 | 4 | 5 | 5 | 4 | 5 | 0 | 0
hours
  Baseline Pre-assessments | 0.603 (0.182) | 0.847 (0.197) | 0.842 (0.333) | 0.762 (0.219) | 0.900 (0.365) | 0.747 (0.220) | 1.079 (0.414) | 0.780 (0.177) |  |
  Baseline Post-assessments: number analyzed (Participants) | 5 | 5 | 4 | 4 | 5 | 4 | 4 | 5 | 0 | 0
  Baseline Post-assessments | 0.357 (0.056) | 0.550 (0.272) | 0.608 (0.431) | 0.242 (0.073) | 0.613 (0.364) | 0.667 (0.426) | 0.562 (0.299) | 0.563 (0.289) |  |
  2-Week Return to School Follow-Up: number analyzed (Participants) | 2 | 4 | 4 | 3 | 2 | 2 | 2 | 3 | 0 | 0
  2-Week Return to School Follow-Up | 1.242 (0.365) | 0.621 (0.138) | 1.208 (0.620) | 0.761 (0.281) | 0.933 (0.094) | 1.133 (0.306) | 1.342 (0.884) | 0.644 (0.287) |  |
  3-Month Return to School Follow-Up: number analyzed (Participants) | 1 | 5 | 3 | 1 | 2 | 2 | 2 | 1 | 0 | 0
  3-Month Return to School Follow-Up | .500 (NA) — n=1 so standard deviation is not relevant | .653 (0.245) | 1.044 (0.474) | 0.250 (NA) — n=1 so standard deviation is not relevant | 0.592 (0.295) | 0.958 (0.295) | 1.017 (0.731) | 0.983 (NA) — n=1 so standard deviation is not relevant |  |

5. Primary Outcome: Average Number of Minutes to Complete Each Intervention Session
Description: Time to complete intervention sessions, each session is expected to last less than 60 minutes. Average calculated by summing all sessions in each condition and dividing by total number of sessions. Note that the number of participants to start a Period is not equal to the number who completed previous Period for "Affect Regulation + Problem Solving" and "Cognitive Restructuring + Problem Solving" because 1 participant in each condition was withdrawn or withdrew.
Time Frame: Baseline
Population: This outcome applies to participants randomized to receive one or more components of the intervention in the Optimization Trial only. Data were not collected for adolescents randomized to the Enhanced Control condition in the Optimization Trial or Hospital Professionals or Adolescent Patients Selected by Hospital Professionals for the Open Trial Period.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Number analyzed (Participants) | 0 | 5 | 6 | 4 | 5 | 5 | 4 | 5 | 0 | 0
minutes |  | 26.864 (12.241) | 26.333 (12.473) | 27.500 (12.103) | 25.938 (13.188) | 37.083 (15.197) | 29.714 (16.838) | 30.522 (14.145) |  |

6. Primary Outcome: Percentage of Adolescent Participants in Which Intervention Delivered With Greater Than or Equal to 80% Fidelity
Description: Percentage of participants in which adherence to delivery of key components of intervention (i.e., skill lessons or practice sessions) across sessions in each condition was 80% or greater. Adherence was calculated based on the number of key components completed relative to the total number of key components expected to be completed for each participant. Note that the number of participants to start a Period is not equal to the number who completed previous Period for "Affect Regulation + Problem Solving" and "Cognitive Restructuring + Problem Solving" because 1 participant in each condition was withdrawn or withdrew.
Time Frame: Baseline
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Number analyzed (Participants) | 0 | 5 | 6 | 4 | 5 | 5 | 4 | 5 | 0 | 0
percentage of participants |  | 100 | 100 | 100 | 100 | 100 | 100 | 100 |  |

7. Primary Outcome: Percentage of Adolescent Participants With Average Acceptability Scores Less Than or Equal to 2
Description: Percent of adolescents with average acceptability score less than or equal to 2 (or "agree") on a five-point scale from 1 (strongly agree) to 5 (strongly disagree). Note that the number of participants to start a Period is not equal to the number who completed previous Period for "Affect Regulation + Problem Solving" and "Cognitive Restructuring + Problem Solving" because 1 participant in each condition was withdrawn or withdrew, and due to missing post-baseline data for "Problem Solving" (1 participant), "Cognitive Restructuring" (1 participant), "Affect Regulation + Cognitive Restructuring" (1 participant), "Cognitive Restructuring + Problem Solving" (1 participant), and "Affect Regulation + Cognitive Restructuring + Problem Solving" (1 participant).
Time Frame: Baseline
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Number analyzed (Participants) | 0 | 5 | 5 | 4 | 4 | 4 | 3 | 4 | 0 | 0
percentage of participants |  | 60 | 60 | 100 | 75 | 50 | 100 | 100 |  |

8. Primary Outcome: Percentage of Hospital Professional Participants With Average Acceptability Scores Less Than or Equal to 2
Description: Percent of hospital professionals with average acceptability score less than or equal to 2 (or "agree") on a five-point scale from 1 (strongly agree) to 5 (strongly disagree). Note that the number of participants to start a Period is not equal to the number who completed previous Period for Hospital Professionals because 7 professionals consented into the study, but only 4 delivered the intervention to a patient following consent.
Time Frame: Baseline
Population: This outcome applies to Hospital Professionals for the Open Trial Period. Data were not collected for adolescents in the Optimization Trial or Adolescent Patients Selected by Hospital Professionals for the Open Trial Period.
Measure: Number; unit: percentage of participants
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
percentage of participants |  |  |  |  |  |  |  |  | 25 |

9. Primary Outcome: Adolescents' Perceptions of Acceptability
Description: Qualitative feedback provided by adolescents receiving the intervention in the Optimization Trial about acceptability of the intervention. Note that the number of participants to start a Period is not equal to the number who completed previous Period for "Affect Regulation + Problem Solving" and "Cognitive Restructuring + Problem Solving" because 1 participant in each condition was withdrawn or withdrew, and due to missing post-baseline data for "Cognitive Restructuring + Problem Solving" (1 participant).
Time Frame: Baseline
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Number analyzed (Participants) | 0 | 5 | 6 | 4 | 5 | 4 | 4 | 5 | 0 | 0
Participants
  Endorsed Part or All of the Intervention |  | 5 | 6 | 4 | 5 | 4 | 4 | 5 |  |
  Identified Aspects that Could Be Improved |  | 5 | 6 | 4 | 5 | 4 | 4 | 5 |  |
  Preferred Learning in Traditional Ways or Described Learning in Virtual Reality as Difficult |  | 1 | 0 | 0 | 0 | 0 | 0 | 1 |  |
  Identified Preference or Benefit to Learning in Virtual Realty (as Opposed to Traditional Ways) |  | 0 | 3 | 0 | 1 | 3 | 1 | 1 |  |

10. Primary Outcome: Hospital Professionals' Perceptions of Acceptability
Description: Qualitative feedback provided by Hospital Professionals delivering the intervention to one or more hospitalized adolescents about acceptability of the intervention. Note that the number of participants to start a Period is not equal to the number who completed previous Period for Hospital Professionals because 7 professionals consented into the study, but only 4 delivered the intervention to a patient following consent.
Time Frame: Baseline
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Participants
  Endorsed Part or All of the Intervention |  |  |  |  |  |  |  |  | 4 |
  Identified Aspects That Could be Improved |  |  |  |  |  |  |  |  | 4 |

ADVERSE EVENTS:
Time Frame: For the Optimization Trial, from signing the informed consent until the 3-Month Return to School Follow-Up or early withdrawal. This time was dependent on the duration of hospital stay and timing of return to school and therefore varied greatly (ranging from 1 day to 405 days). For the Open Trial Period, adverse events for the Adolescent Patients Selected by Hospital Professionals were only monitored during intervention delivery.
Description: The Open Trial Period Hospital Professionals were not considered to be at risk for adverse events and data were not collected for this arm.
Arm/Group | Enhanced Control | Affect Regulation | Problem Solving | Affect Regulation + Problem Solving | Cognitive Restructuring | Affect Regulation + Cognitive Restructuring | Cognitive Restructuring + Problem Solving | Affect Regulation + Cognitive Restructuring + Problem Solving | Hospital Professionals | Adolescent Patients Selected by Hospital Professionals
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/6 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/0 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/5 | 1/6 | 1/5 | 1/5 | 1/5 | 0/5 | 3/5 | 0/0 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 1/5 | 0/6 | 0/5 | 0/5 | 0/5 | 0/5 | 1/5 | 0/0 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Control (N=6) | Affect Regulation (N=5) | Problem Solving (N=6) | Affect Regulation + Problem Solving (N=5) | Cognitive Restructuring (N=5) | Affect Regulation + Cognitive Restructuring (N=5) | Cognitive Restructuring + Problem Solving (N=5) | Affect Regulation + Cognitive Restructuring + Problem Solving (N=5) | Hospital Professionals (N=0) | Adolescent Patients Selected by Hospital Professionals (N=5)
Emergency Department Visit for Suicide-Related Risk or Associated Symptoms (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Hospitalization for Suicide-Related Risk or Associated Symptoms (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hospitalization for Medical Procedure: GI (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hospitalization for Medical Procedure: Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parent Distress Related to Adolescent Risk Behaviors (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Parent concern related to adolescent psychiatric concerns (i.e., suicide-related risk and running away)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Control (N=6) | Affect Regulation (N=5) | Problem Solving (N=6) | Affect Regulation + Problem Solving (N=5) | Cognitive Restructuring (N=5) | Affect Regulation + Cognitive Restructuring (N=5) | Cognitive Restructuring + Problem Solving (N=5) | Affect Regulation + Cognitive Restructuring + Problem Solving (N=5) | Hospital Professionals (N=0) | Adolescent Patients Selected by Hospital Professionals (N=5)
Distress (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical Procedure or Action (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Evaluated for ingesting a coin
Medical Action (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Assessment of syncope symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT05934396/Prot_SAP_001.pdf
  • Informed Consent Form (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT05934396/ICF_000.pdf